CLINICAL TRIAL: NCT05834140
Title: Effects of Muscle Energy Technique on Post-Dural Puncture Headache, Neck Pain and Disability After Cesarean Section
Brief Title: Effects of MET on PPDH, Neck Pain and Disability After Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0510
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Post-Dural Puncture Headache; Cesarean Section Complications
Keywords: post dural puncture headache; neck pain; Cesarean Section
MeSH Terms: conditions — Post-Dural Puncture Headache; Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional physical therapy (Active Comparator): TENS and Heating pads
  Interventions: Other: Traditional Physical Therapy
- Muscle Energy Technique (Experimental): Muscle Energy Technique protocol in along with TENS and Heating pads
  Interventions: Other: Muscle Energy Technique

INTERVENTIONS:
Other: Traditional Physical Therapy — TENS (transcutaneous electrical nerve stimulation) on continuous mode at 80-120 Hz for 15-20 min and Heating pads for 10-15 min
  Total 4 sessions will be given in 2 days
  Arms: Traditional physical therapy
Other: Muscle Energy Technique — Muscle energy technique (Post Isometric relaxation) along with TENS and Heating pads.
  * MET of the scaleni
  * MET of Sternocleidomastoid
  * MET of Levator Scapulae
  * MET of Upper fibers of Trapezius
  Total 4 sessions will be given in 2 days
  Arms: Muscle Energy Technique

SUMMARY:
The goal of this clinical trial is to determine the effect of Muscle Energy Techniques on post dural puncture headache, neck pain and disability after Cesarean Section.

.

DETAILED DESCRIPTION:
Caesarean section (CS) is the worldwide process of pregnancy termination that delivers live or dead fetuses with an incision on the abdominal wall and uterine wall.

It is performed under neuraxial anesthesia (spinal and epidural anesthesia). Post- dural puncture headache (PDPH) is a major complication of neuraxial anesthesia which presents as a dull throbbing pain in a frontal-occipital distribution, aggravates on sitting or standing, and is reduced by lying down.

This study will be a randomized clinical trial. Subjects with PPDH meeting the predetermined inclusion and exclusion criteria will be divided into two groups: i.e. treatment and control group. Both groups will receive baseline treatments i.e. (heating pads & TENS). In addition, treatment group will receive post-isometric relaxation of METs. Each subject will receive a total of 4 treatment sessions, with 2 treatment sessions per day

Pre-treatment will be done at day 1 and post-treatment will be done at day 2, using Headache Disability Index (HDI), Numeric Pain Rating Scale (NPRS) and Neck Disability Index (NDI) as subjective measurements. Recorded values will be analysed for any change using SPSs

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 40 years
* Both Primiparous and multiparous
* Both elective and emergency Lower Section Cesarean Section
* Headache occurring within 24-72 hours post C-section
* Headache aggravates on getting in upright position

Exclusion Criteria:

* History of Trauma/fracture of head and neck region
* History of cervical spine surgery
* Had previous diagnostic Lumbar Puncture (LP)
* Any kind of infection, malignancy, inflammation and structural deformity present in head and neck region.
* Other serious forms of headaches including Migraine, Cluster, thunderclap, hypnic etc.
* Cervical Radiculopathies and spondylolisthesis

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 2nd day
  Numeric pain rating scale (NPRS) is an outcome measure that is a segmented numeric version of visual analogue scale in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of patient's pain. The common format is horizontal bar or line and NPRS is anchored by terms describing pain and severity extremes
Neck Disability Index | 2nd day
  The NDI is a 10-item scaled self-administered questionnaire covering pain, concentration, and activities of daily living. Each of the ten items is scored from 0 to 5, and the total is calculated and multiplied by two to produce a percentage score of the maximal score; higher score indicates greater disability. Vernon and Mior defined 0-8 as none, 10-28 as mild, 30-48 as moderate, 50-68 as severe, and over 68 as complete disability
Headache Disability Index | 2nd day
  The Henry Ford Hospital Headache Disability Questionnaire (HDI) is a 25-item questionnaire that examines the effects of headache on daily life. This questionnaire has a two-factor structure emotionally and functionally. Scoring (No: 0, Sometimes:2, Yes:4) varies between 0 and 100. The higher the score, the more headache disability

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam Muneeb, MPhil, Principal Investigator — Riphah International University
Locations (1):
- Madinah Teaching Hospital, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwak KH. Postdural puncture headache. Korean J Anesthesiol. 2017 Apr;70(2):136-143. doi: 10.4097/kjae.2017.70.2.136. Epub 2017 Feb 3. PMID 28367283
- [Background] Halalmeh DR, Sandio A, Adrian M, Moisi MD. Intracranial Subdural Hematoma Versus Postdural Puncture Headache Following Epidural Anesthesia: A Case Report. Cureus. 2022 Feb 1;14(2):e21824. doi: 10.7759/cureus.21824. eCollection 2022 Feb. PMID 35291537
- [Background] Patel R, Urits I, Orhurhu V, Orhurhu MS, Peck J, Ohuabunwa E, Sikorski A, Mehrabani A, Manchikanti L, Kaye AD, Kaye RJ, Helmstetter JA, Viswanath O. A Comprehensive Update on the Treatment and Management of Postdural Puncture Headache. Curr Pain Headache Rep. 2020 Apr 22;24(6):24. doi: 10.1007/s11916-020-00860-0. PMID 32323013
- [Background] Yang XJ, Sun SS. Comparison of maternal and fetal complications in elective and emergency cesarean section: a systematic review and meta-analysis. Arch Gynecol Obstet. 2017 Sep;296(3):503-512. doi: 10.1007/s00404-017-4445-2. Epub 2017 Jul 5. PMID 28681107
- [Background] Segraves RL, Segraves JM. Reducing Maternal Morbidity on the Frontline: Acute Care Physical Therapy After Cesarean Section During and Beyond the COVID-19 Pandemic. Phys Ther. 2021 Jul 1;101(7):pzab093. doi: 10.1093/ptj/pzab093. No abstract available. PMID 33713410
- [Background] Kato S, Takeshita K, Matsudaira K, Tonosu J, Hara N, Chikuda H. Normative score and cut-off value of the Neck Disability Index. J Orthop Sci. 2012 Nov;17(6):687-93. doi: 10.1007/s00776-012-0276-y. Epub 2012 Aug 16. PMID 22895822